CLINICAL TRIAL: NCT03382899
Title: A Randomized Phase 2 Trial of AM0010 in Combination With Pembrolizumab vs. Pembrolizumab Alone as First-Line (1L) Therapy in Patients With Stage IV / Metastatic Wild Type (WT) Non-Small Cell Lung Cancer and Tumors With High Expression of PD-L1 (> 50%)
Brief Title: Study of Pegilodecakin (LY3500518) With Pembrolizumab Compared to Pembrolizumab Alone First-line Tx in Participants With Metastatic Non-Small Cell Lung Cancer
Acronym: Cypress 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The CYPRESS-1 trial was closed early after the planned primary analysis because the risk benefit ratio is unfavorable.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17160; J1L-AM-JZGC (Other: Eli Lilly and Company); AM0010-201 (Other: ARMO BioSciences)
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pegilodecakin; AM0010; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegilodecakin + Pembrolizumab (Experimental): Participants received pegilodecakin subcutaneously (SQ) at 0.8 milligrams (mg) (≤80 kilograms (kg) body weight) or 1.6 mg (>80 kg body weight) once daily (QD) in the abdomen, thigh or back of upper arm.
  Pembrolizumab administered as an intravenous (IV) infusion at 200 mg on Day 1 of a 21-day cycle.
  Interventions: Biological: Pegilodecakin; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): Participants received pembrolizumab as an IV infusion at 200 mg on Day 1 of a 21-day cycle.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Biological: Pegilodecakin — Pegilodecakin plus Pembrolizumab
  Other Names: LY3500518; AM0010
  Arms: Pegilodecakin + Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab Alone

SUMMARY:
To compare the efficacy of pegilodecakin in combination with pembrolizumab versus pembrolizumab alone in participants with metastatic non-small cell lung cancer as measured by objective response rate.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized, Phase 2 study designed to compare the efficacy and safety of pegilodecakin in combination with pembrolizumab versus pembrolizumab alone in participants with stage IV / metastatic wild type non-small cell lung cancer and tumors with high expression of PD-L1 (> 50%).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed WT NSCLC that is stage IV / metastatic or recurrent
2. Participants with tumor tissue high expression of PD-L1 as defined by Tumor Proportion Score (TPS) ≥ 50%
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Participants with measurable disease by spiral CT or MRI per RECIST v.1.1 criteria.
5. Participants that have completed prior radiotherapy or radiosurgery at least 2 weeks prior to randomization.
6. Participants must be naïve to therapy for the advanced stage of the disease. Previous neoadjuvant or adjuvant therapy is allowed for participants who successfully underwent complete radical surgery and ONLY if the last treatment was administered more than 12 months prior to the start of the trial treatment

Exclusion Criteria:

1. Participants with active central nervous system (CNS) metastases or carcinomatous meningitis
2. Participants with any serious or uncontrolled medical disorder or active infection with the hepatitis virus or the human immunodeficiency virus (HIV)
3. Participants with Grade 1 (NCI-CTCAE v.4.03) toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue prior to randomization
4. Participants that have received pembrolizumab
5. Participants with a history of severe hypersensitivity reactions to monoclonal antibodies
6. Pregnant or lactating women
7. Participants receiving any investigational agent within 28 days of first administration of trial treatment
8. Participants that have received therapy with anti-tumor vaccines or other immunostimulatory antitumor agents
9. Participants that have received therapy with anti-PD-1, anti-PD-L1, anti-PD-L-2, anti-CD-137, and/or anti CTLA-4 antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (74):
  - CCI - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Oncology Associates, P.C., Tempe, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - St. Joseph Heritage Medical Group, Fullerton, California
  - Glendale Adventist Medical Center, Los Angeles, California
  - Redlands Community Hospital, Redlands, California
  - Redwood Regional Oncology Center, Santa Rosa, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Kaiser Permanente Oncology Clinic, Denver, Colorado
  - Rocky Mountain Cancer Center, Lone Tree, Colorado
  - Veterans Affairs Connecticut Healthcare System, West Haven, Connecticut
  - Medical Oncology Hematolgy Consultants, PA, Newark, Delaware
  - Lynn Cancer Institute Ctr for Hem-Onc, Boca Raton, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - SCRI- Florida Cancer Specialists, Tallahassee, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - AMITA Health Cancer Institute & Outpatient Center, Hinsdale, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Goshen Health System, Goshen, Indiana
  - University of Iowa, Iowa City, Iowa
  - Covenant Clinic, Waterloo, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Baptist Health Medical Group, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - MedStar Research Institute, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital Detroit, Detroit, Michigan
  - Sparrow Health System, Lansing, Michigan
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - St John's Mercy Medical Center, St Louis, Missouri
  - Nebraska Hematology-Oncology, Lincoln, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - The Valley Hospital - Luckow Pavilion, Westwood, New Jersey
  - Clinical Research Alliance, Inc., Lake Success, New York
  - Winthrop University Hospital, Mineola, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Jacksonville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - The Toledo Clinic, Toledo, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Texas Cancer Center (Abilene), Abilene, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Texas Oncology - Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - US Oncology, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology-Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology-Wichital Falls Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax Northern Virginia Hematology Oncology, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Roanoke, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
  - MultiCare Regional Cancer Center - Auburn, Tacoma, Washington
  - The Richland Hospital, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Spigel D, Jotte R, Nemunaitis J, Shum M, Schneider J, Goldschmidt J, Eisenstein J, Berz D, Seneviratne L, Socoteanu M, Bhanderi V, Konduri K, Xia M, Wang H, Hozak RR, Gueorguieva I, Ferry D, Gandhi L, Chao BH, Rybkin I. Randomized Phase 2 Studies of Checkpoint Inhibitors Alone or in Combination With Pegilodecakin in Patients With Metastatic NSCLC (CYPRESS 1 and CYPRESS 2). J Thorac Oncol. 2021 Feb;16(2):327-333. doi: 10.1016/j.jtho.2020.10.001. Epub 2020 Nov 6. PMID 33166722

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that had a recorded death on study or are alive and being followed at the end of the trial but off treatment are considered as completed group
Period: Overall Study
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Started | 51 | 50
Received at Least 1 Dose of Study Drug | 50 | 48
Completed | 20 | 15
Not Completed | 31 | 35
Not completed — Ineligibility Determined | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor's decision | 31 | 28
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Pegilodecakin + Pembrolizumab: Participants received pegilodecakin SQ at 0.8 mg (≤80 kg body weight) or 1.6 mg (>80 kg body weight) QD in the abdomen, thigh or back of upper arm.
  Pembrolizumab administered as an IV infusion at 200 mg on Day 1 of a 21-day cycle.
- Pebrolizumab: Participants received pembrolizumab as an IV infusion at 200 mg on Day 1 of a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Pegilodecakin + Pembrolizumab | Pebrolizumab | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (7.7) | 67.1 (9.0) | 67.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 28 | 32 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 40 | 47 | 87
  Unknown or Not Reported | 8 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 39 | 38 | 77
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Objective Response Rate (ORR)
Description: ORR defined as the percentage of participants who achieve a CR or PR as assessed by RECIST v.1.1. The ORR is the number of participants with a complete response (CR) or partial response (PR) divided by the number of randomized participants recorded between the date of randomization and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever comes first. Complete response (CR) is defined as disappearance of all target (and non-target) lesions, and normalization of tumor marker level. Partial response (PR) is defined as at least a 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: From Date of Randomization to Progressive Disease, Death from Any cause (Up to 24 Months)
Population: All randomized participants who had adequate baseline and at least 1 post-baseline tumor assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 51 | 50
percentage of participants | 47.1 [32.9 to 61.5] | 44.0 [30.0 to 58.8]
Statistical Analysis 1: Comparison: Pegilodecakin + Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.7626, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.5 to 2.5] — Odds Ratio stratified by histology type, squamous versus non-squamous based on interactive web response system (IWRS). 95% Confidence intervals (CIs) were estimated using the Clopper-Pearson method

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to death due to any cause. Participants who were alive at the end of the follow-up period or lost to follow-up were censored on the last date the participant was known to be alive.
Time Frame: From Date of Randomization to Death Due to Any Cause (Up to 24 Months)
Population: All randomized participants. Censored participants in the Pegilodecakin + Pembrolizumab arm is 32 and the Pembrolizumab arm is 39.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 51 | 50
Months | 16.33 [10.51 to NA] — The upper 95% confidence interval was not achieved due to high censoring rate. | NA [NA to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate.
Statistical Analysis 1: Comparison: Pegilodecakin + Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.263, Log Rank; Hazard Ratio (HR) = 1.530, 95% CI 2-sided [0.722 to 3.243] — Hazard Ratio stratified by histology type, squamous versus non-squamous based on IWRS. 95% CIs were estimated using the methods of Brookmeyer and Crowley, and Greenwood, respectively

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of randomization to the earlier of first documentation of disease progression or death due to any cause. Progressive disease (PD) is defined by at least a 20% increase in the sum of longest diameters of target lesions, taking as reference the baseline sum of longest diameters or the presence of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression determined by scans. Participants who did not progress, who discontinued treatment for toxicity or a reason other than documented progression, or who were lost to follow up before documented progression and death or were censored at the date of last adequate tumor assessment, participants or new anticancer therapy started and not tumor progression or death were censored at the last adequate tumor assessment before the start of new anticancer therapy.
Time Frame: From Date of Randomization to Progressive Disease (PD) or Death Due to Any Cause (Up to 24 Months)
Population: All randomized participants. Censored participants in the Pegilodecakin + Pembrolizumab arm is 24 and Pembrolizumab arm is 22.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 51 | 50
Months | 6.28 [2.86 to NA] — Upper limit of confidence interval was not reached. | 6.08 [2.23 to NA] — Upper limit of confidence interval was not reached.
Statistical Analysis 1: Comparison: Pegilodecakin + Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.20, Log Rank; Hazard Ratio (HR) = 0.975, 95% CI 2-sided [0.571 to 1.663] — Hazard Ratio stratified by histology type, squamous versus non-squamous based on IWRS. 95% CIs were estimated using the Kaplan-Meier method

4. Secondary Outcome: Percentage of Participants Who Achieved a Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants in the analysis population who have achieved a complete response (CR), partial response (PR) or stable disease (SD) response prior to disease progression. CR is defined as disappearance of all target (and non-target) lesions, and normalization of tumor marker level. PR is defined as at least a 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of longest diameters. SD is defined as neither sufficient shrinkage of target lesions to qualify for partial response, nor sufficient increase to qualify for progressive disease, taking as reference the baseline sum of longest diameters.
Time Frame: From Date of Randomization to Objective Progressive Disease or Start of New Anti-Cancer Therapy (Up to 24 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 51 | 50
percentage of participants | 62.7 [48.1 to 75.9] | 62.0 [47.2 to 75.4]
Statistical Analysis 1: Comparison: Pegilodecakin + Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.9418, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.5 to 2.3] — Odds Ratio stratified by histology type, squamous versus non-squamous based on IWRS. 95% CIs were estimated using the Clopper-Pearson method

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the earliest date of qualifying response until earliest date of disease progression per RECIST v1.1 or death from any cause, whichever comes first. Duration of response was analyzed in participants who had CR or PR. Duration of response was censored on the date of the last tumor assessment on trial for participants who did not have objective tumor progression and who did not die due to any cause while on trial. For participants who discontinued participation in the trial or discontinued from tumor scan assessments before disease progression, the duration of response was censored at the date of the last tumor assessment.
Time Frame: From Date of Response to Death Due to Any Cause (Up to 24 Months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 51 | 50
Months | 14.23 [2.50 to 14.23] | NA [4.14 to NA] — Median was not calculated and upper limit confidence interval was not reached.
Statistical Analysis 1: Comparison: Pegilodecakin + Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.8312, Log Rank; Hazard Ratio (HR) = 1.124, 95% CI 2-sided [0.384 to 3.289] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline Up To 24 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Pegilodecakin + Pembrolizumab | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 19/50 | 13/48
Serious Adverse Events (participants affected / at risk) | 28/50 | 25/48
Other Adverse Events (participants affected / at risk) | 48/50 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegilodecakin + Pembrolizumab (N=50) | Pembrolizumab (N=48)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 6 (6)
Sepsis (Infections and infestations) | 5 (6) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Capillary leak syndrome (Vascular disorders) | 1 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pegilodecakin + Pembrolizumab (N=50) | Pembrolizumab (N=48)
Anaemia (Blood and lymphatic system disorders) | 30 (92) | 10 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (28) | 5 (9)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (4)
Constipation (Gastrointestinal disorders) | 5 (6) | 16 (19)
Diarrhoea (Gastrointestinal disorders) | 12 (23) | 11 (16)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 14 (16) | 10 (12)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (7)
Asthenia (General disorders) | 4 (4) | 3 (3)
Chills (General disorders) | 7 (8) | 1 (2)
Fatigue (General disorders) | 27 (41) | 23 (25)
Injection site reaction (General disorders) | 4 (5) | 2 (3)
Localised oedema (General disorders) | 1 (1) | 3 (3)
Malaise (General disorders) | 1 (6) | 3 (3)
Non-cardiac chest pain (General disorders) | 5 (6) | 1 (1)
Oedema peripheral (General disorders) | 9 (9) | 10 (12)
Pyrexia (General disorders) | 13 (16) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (6) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 7 (9) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (9) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 5 (8) | 4 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (5) | 1 (4)
Blood creatinine increased (Investigations) | 6 (15) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 6 (13) | 4 (9)
Weight decreased (Investigations) | 5 (6) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 19 (21) | 16 (16)
Dehydration (Metabolism and nutrition disorders) | 11 (12) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (15) | 11 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (12) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Dizziness (Nervous system disorders) | 7 (8) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 6 (10)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (3)
Depression (Psychiatric disorders) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (9) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/22 (0) | 1/18 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 13 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (28) | 13 (24)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 13 (21) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (12)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 13 (17) | 3 (8)

LIMITATIONS AND CAVEATS:
Study was terminated early after completion of primary analysis; hence, no mature data were available for final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03382899/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03382899/SAP_001.pdf